CLINICAL TRIAL: NCT04072120
Title: Stroke Survival in Municipalities: Impact of Geographic Proximity to First- and Second-degree Relatives
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oslo (Other)
Collaborators: Extrastiftelsen (Other); The National Association for Public Health, Norway (Other Government)
Responsible Party: Principal Investigator, CHOI, HYE JUNG, Doctoral Research Fellow, University of Oslo
Other Study IDs: NorStrokeSurvival
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Stroke
Keywords: Stroke; Post-acute stroke; Geographical proximity; Family; Relatives; Survival analysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- R1: 1. Norwegian citizens aged 45 and above 1.1.1994 - 31.12. 2009 registered in the FS-data during this period.
  2. Sub-sample those attending a cardiovascular health survey who later developed stroke.
- R2: All Norwegians born in the period 1 January 1940 to 31 December 1959 who survived to 1991.
- R3: Norwegian citizens aged 45 and above 1.1.2016.

SUMMARY:
Our key objective will be to investigate if geographic proximity to first- and second-degree relatives has an influence on post-acute stroke survival and use of health and social services. We will also model and map spatial variation in stroke and cardiovascular disease (CVD) incidence and mortality and see if some of the variation is due to spatial clustering of familial risk. The study will use innovative approaches to large-scale registry and survey data and statistical analysis on the full Norwegian population. We will integrate multigenerational and geographical information. This will enable us to assess key determinants on stroke survival and use of health and social care at municipality level.

ELIGIBILITY:
Inclusion Criteria:

* Norwegian citizens aged 45 and above 1.1.1994 - 31.12. 2009 and had stroke events
* Those who attend a cardiovascular health survey who later developed stroke.
* All Norwegians born in the period 1 January 1940 to 31 December 1959 who survived to 1991
* Norwegian citizens aged 45 and above 1.1.2016 and had stroke events

Exclusion Criteria:

-

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. All Norwegian residents in the period from 1960 to 2017 (n=7,4 mill), including all births and deaths(from the Cause of Death Registry) occurring in this population from 1960 onwards.
  2. The Multigenerational Register in Statistics Norway covering family linkage on all individuals to their parents for all born after 1952 is included.
  3. The Census from 1960, and from 1970 to 2011
  4. Hospital data on hospital discharge from cardiovascular events among all Norwegians from 1992.
Sampling Method: Non-Probability Sample
Enrollment: 7400000 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-08-14 (Estimated); Study Completion 2022-08-14 (Estimated)

PRIMARY OUTCOMES:
R1- Mortality | Mortality follow-up from 1.1.1994 to 31.12.2014
  Mortality of Norwegian citizens aged 45 and above 1.1.1994 - 31.12. 2009
R2- Mortality | Mortality follow-up from 1991-2014.
  Mortality of all Norwegians born in the period 1 January 1940 to 31 December 1959 who survived to 1991
R3- Stroke events | Stroke events registered in the Patient registry after 2016, (possibly until 2019)
  Norwegian citizens aged 45 and above 1.1.2016

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Næss, MD, MSc, PhD, Principal Investigator — Department of Community Medicine and Global Health, University of Oslo
Locations (1):
- Department of Community Medicine and Global Health,University of Oslo, Oslo, Norway